CLINICAL TRIAL: NCT03419026
Title: Pregnant Exposure to Persistent Organic Pollutants With Endocrine Disrupting Activity and Development of Breast Cancer in the Next 15 Years: Longitudinal Prospective Cohort Nested Case-control Study
Brief Title: Pregnant Exposure to Persistent Organic Pollutants
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 16AOI10
Record Dates: First submitted 2017-11-20; First posted 2018-02-01 (Actual); Last update posted 2018-02-01 (Actual); Status verified 2017-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- breast cancer
- control

SUMMARY:
Breast cancer, the first female cancer, affects one in eight women in her lifetime. The increase and uneven distribution of its prevalence throughout the world cannot be fully explained either by the increase in life expectancy, or by genetic factors present in less than 10% of cases, or by early detection, or by the use of hormone therapy for menopause at certain periods of time.

Numerous experimental and epidemiological arguments, as well as the increased risk of breast cancer in women after 50 years of age who were exposed in utero to Distilbene prescribed for their mothers in the 1950s to 75's, suggest the involvement of environmental factors involved in early development (nutrition, alcohol, tobacco, chemical pollutants) that may act as endocrine disruptors, estrogenomimetic or intervening on other nuclear receptors such as the However, the formal demonstration of the deleterious physiopathological role of such exposure comes up against methodological difficulties in epidemiological terms: first of all, the fact that correlation is sought at the time of the discovery of breast cancer when there are critical windows of exposure (fetal, perinatal, peripubertal and pregnant) and that persistent organic products or POPs, most often lipids, are present.

The objective of this project is to correlate the per-gravidic exposure to POPs (dioxins, dioxinlike, polychlorinated bisphenyls, organochlorine pesticides and flame-retardant polybrominated derivatives) and the development, within 15 years of delivery, of breast cancer, taking into account the confounding factors of classical breast cancer risk (age, reproductive events, etc.).

This project benefits on the one hand from a cord blood bank set up between 2002 and 2005 (6,242 samples) carried out at the Nice University Hospital and the Grasse University Hospital, during a PHRC and on the other hand from the cancer observatory / CRISAP of the PACA Corsica region, exhaustive to more than 92% since 2005, registers which will be cross-referenced and whose cancer cases (N) will be compared to controls. The assays will be carried out after purification, using high-resolution mass spectrometry gas chromatography coupling, the quantification being carried out according to the principle of isotopic dilution. They will be carried out by LABERCA in Nantes, the national reference laboratory of the French Health Agencies ANSES and INVS and also involved in various European projects. Concentrations related to blood lipids will be expressed in quartile and analyzed separately or combined with a cumulative score taking into account confounding risk factors for breast cancer and the geolocation of the initial and final residence in relation to the incinerator of the City of Nice (Department of Public Health CHU of Nice).

DETAILED DESCRIPTION:
Breast cancer, the first female cancer, affects one in eight women in her lifetime. The increase and uneven distribution of its prevalence throughout the world cannot be fully explained either by the increase in life expectancy, or by genetic factors present in less than 10% of cases, or by early detection, or by the use of hormone therapy for menopause at certain periods of time.

Numerous experimental and epidemiological arguments, as well as the increased risk of breast cancer in women after 50 years of age who were exposed in utero to Distilbene prescribed for their mothers in the 1950s to 75's, suggest the involvement of environmental factors involved in early development (nutrition, alcohol, tobacco, chemical pollutants) that may act as endocrine disruptors, estrogenomimetic or intervening on other nuclear receptors such as the However, the formal demonstration of the deleterious physiopathological role of such exposure comes up against methodological difficulties in epidemiological terms: first of all, the fact that correlation is sought at the time of the discovery of breast cancer when there are critical windows of exposure (fetal, perinatal, peripubertal and pregnant) and that persistent organic products or POPs, most often lipids, are present.

The objective of this project is to correlate the per-gravidic exposure to POPs (dioxins, dioxinlike, polychlorinated bisphenyls, organochlorine pesticides and flame-retardant polybrominated derivatives) and the development, within 15 years of delivery, of breast cancer, taking into account the confounding factors of classical breast cancer risk (age, reproductive events, etc.).

This project benefits on the one hand from a cord blood bank set up between 2002 and 2005 (6,242 samples) carried out at the Nice University Hospital and the Grasse University Hospital, during a PHRC and on the other hand from the cancer observatory / CRISAP of the PACA Corsica region, exhaustive to more than 92% since 2005, registers which will be cross-referenced and whose cancer cases (N) will be compared to controls. The assays will be carried out after purification, using high-resolution mass spectrometry gas chromatography coupling, the quantification being carried out according to the principle of isotopic dilution. They will be carried out by LABERCA in Nantes, the national reference laboratory of the French Health Agencies ANSES and INVS and also involved in various European projects. Concentrations related to blood lipids will be expressed in quartile and analyzed separately or combined with a cumulative score taking into account confounding risk factors for breast cancer and the geolocation of the initial and final residence in relation to the incinerator of the City of Nice (Department of Public Health CHU of Nice).

The implementation of such a protocol requires a preliminary feasibility phase, which is the subject of this AOI request and which will depend on:

1. Sending a letter to the 6242 mothers whose sera (derived from cord blood) are stored in the bank set up between 2002 and 2005 in order to

   1. Verify that they still live in the PACA region
   2. confirm their willingness to participate in this study on the exposure/emergence relationship of breast cancer by serum assay.

   (c) indicate whether they agree to be part of the follow-up cohort
2. Determination, by crossing the two registers (cord blood bank) and cancer register / CRISAP, of women who gave birth at the Nice University Hospital or at the Grasse University Hospital of a boy between 2002 and 2005 and who developed breast cancer in the next 13 years (considered N cases); who have not developed breast cancer and will be matched for age and date of delivery (controls 2N).
3. Determination of their gynaecological characteristics, breast cancer risk factors and cancer characteristics.

The project will then continue beyond the AOI, through the determination of dioxins, dioxins-like, PCBs and brominated derivatives in the context of specific funding, and the analysis of results.

These privileged conditions should make it possible, by resolving some of the methodological difficulties inherent in the environmental epidemiology of cancers, to provide information on the possible role of exposure to persistent organic products during critical periods, such as pregnancy in the occurrence of breast cancer, and to justify preventive measures and the development of new predictive risk factors.

ELIGIBILITY:
Inclusion Criteria:

woman who gave birth between 2002 and 2005 to a boy whose cord blood was stored in a 2002/2005 PHRC.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: woman who gave birth between 2002 and 2005 to a boy whose cord blood was stored in a 2002/2005 PHRC.
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
the Number of blood samples usable by return of patient non-opposition | 1 year
  To make it possible from a regulatory and ethical point of view to use the exceptional bank of 6242 cord blood samples collected between 2002 and 2005 in the Nice (CHU) and Grasse maternity hospitals (CHR) and stored in the biochemistry laboratory (CHU Nice) in order to seek an association between the per-gravidic exposure to the main persistent organic pollutants of dioxins or dioxins-like type and the early onset in pregnant women.

CONTACTS AND LOCATIONS:
Locations (1):
- Nice Hospital, Nice, France

IPD SHARING:
Plan to Share IPD: No